CLINICAL TRIAL: NCT04305379
Title: Augmented BLAdder NecK rEconstruction Trial for Improved Urinary Function After Radical Prostatectomy
Acronym: BLANKET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped due to COVID-19 pandemic, low priority among initiatives and officially terminated.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00208651
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer; Urinary Incontinence; Surgery
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The surgeon will be masked until the time of bladder neck reconstruction during the radical prostatectomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Bladder Neck Reconstruction (Experimental): Augmented Bladder Neck Reconstruction (Sling + Intussusception)
  Interventions: Procedure: Augmented Bladder Neck Reconstruction
- Standard Bladder Neck Reconstruction (Active Comparator): Standard Bladder Neck Reconstruction (Intussusception Only)
  Interventions: Procedure: Standard Bladder Neck Reconstruction

INTERVENTIONS:
Procedure: Augmented Bladder Neck Reconstruction — Augmented Bladder Neck Reconstruction including a Medial Umbilical Ligament Sling plus Intussusception
  Arms: Augmented Bladder Neck Reconstruction
Procedure: Standard Bladder Neck Reconstruction — Standard Bladder Neck Reconstruction with Intussusception Only
  Arms: Standard Bladder Neck Reconstruction

SUMMARY:
The investigators are conducting a prospective, randomized trial to investigate whether patients randomized to receive an augmented bladder neck reconstruction (aBNR) at the time of robotic-assisted laparoscopic prostatectomy experience improved urinary function post-operatively compared to patients who undergo prostatectomy with a standard BNR. An aBNR here consists of the autologous medial umbilical ligament sling as well as a bladder neck intussusception stitch. The standard BNR group will receive the intussusception stitch only.

DETAILED DESCRIPTION:
A bladder neck reconstruction is a standard step in performing a radical prostatectomy. Over the years, various maneuvers to improve continence have been tried and studied including intussusception stitches and slings. Slings of various origins have been used by surgeons at the time of radical prostatectomy without consistent evidence demonstrating a benefit (vas deferens, biologic). However, use of the medial umbilical ligament to create a sling has not previously been studied in a randomized trial.

The medial umbilical ligaments are normally cut during intraperitoneal robotic-assisted laparoscopic radical prostatectomy to allow the surgeon access to the Retzius space between the bladder and pubic bone. To create a medial umbilical ligament autologous sling, the ligaments are dissected out and wrapped around the vesicourethral anastomosis.

The investigators are conducting a prospective, randomized trial to investigate whether patients randomized to receive an augmented bladder neck reconstruction (aBNR) at the time of robotic-assisted laparoscopic prostatectomy experience improved urinary function post-operatively compared to patients who undergo prostatectomy with a standard BNR. An aBNR here consists of the autologous medial umbilical ligament sling as well as a bladder neck intussusception stitch. The standard BNR group will receive the intussusception stitch only.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 40 to 70 years of age with localized prostate cancer (clinical stage T2c or less, Gleason grade 5+5=10 or less without any evidence of distant metastases)
* Scheduled to undergo curative robot-assisted radical prostatectomy

Exclusion Criteria:

* Planned pre-operative or post-operative (within 1 month) androgen therapy
* Planned pre-operative or post-operative (within 1 month) radiation therapy
* History of spinal trauma or surgery to the brain or spinal cord
* Pre-operative history of stress urinary incontinence

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
EPIC Urinary Incontinence subscale score | 1 Month
  Score of 0-100 on questionnaire with higher scores reflecting better health-related quality of life related to urinary incontinence (closer to 0 is more incontinence, closer to 100 is less incontinence).

SECONDARY OUTCOMES:
EPIC Urinary Incontinence subscale score | 2 Weeks
  Score of 0-100 on questionnaire with higher scores reflecting better health-related quality of life related to urinary incontinence (closer to 0 is more incontinence, closer to 100 is less incontinence).
EPIC Urinary Incontinence subscale score | 3 Months
  Score of 0-100 on questionnaire with higher scores reflecting better health-related quality of life related to urinary incontinence (closer to 0 is more incontinence, closer to 100 is less incontinence).
EPIC Urinary Incontinence subscale score | 6 Months
  Score of 0-100 on questionnaire with higher scores reflecting better health-related quality of life related to urinary incontinence (closer to 0 is more incontinence, closer to 100 is less incontinence).
EPIC Urinary Incontinence subscale score | 12 Months
  Score of 0-100 on questionnaire with higher scores reflecting better health-related quality of life related to urinary incontinence (closer to 0 is more incontinence, closer to 100 is less incontinence).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad E Allaf, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No